CLINICAL TRIAL: NCT04902209
Title: Static Balance Disorders in Patients After ( (ORIF) Surgical Treatment of Hip Acetabular Fractures
Brief Title: Static Balance Disorders in Patients After Surgical Treatment of Hip Acetabular Fractures
Status: Completed | Type: Observational
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: Ds 310/SN4
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Hip Fractures; Acetabular Fracture; Balance; Distorted; Disability Physical
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1- study group- patients after surgical treatment of acetabular fracture: 1- study group- patients after surgical treatment of hip acetabular fracture
  Interventions: Procedure: postural stability measurements
- 2- control group- healthy subjects: 2- control group- healthy subjects age, BMI matched
  Interventions: Procedure: postural stability measurements

INTERVENTIONS:
Procedure: postural stability measurements — Static balance assessment on bi-module stabilometric platform CQStab2P. It registers the movement of centre of foot pressure (COP).
  Harris hip score- disability assesment
  Other Names: harris hip score

SUMMARY:
The mechanism of maintaining balance is a complex phenomenon, involving numerous systems of human body. High-energy trauma resulting in acetabular fracture damages some of the elements composing this delicate mechanism, potentially increasing the risk of falls in patients. There have not been any studies so far on balance levels in patients after surgical treatment of acetabular fractures.

Questions/purposes

1. Do balance disorders occur in patients after ORIF of acetabular fractures?
2. Do surgical approach and fracture pattern influence balance level of patients?
3. Should therapy programs include certain stabilometric parameters adequate especially for this type of injury?

DETAILED DESCRIPTION:
Methods Between 2014-2017, investigators evaluated 110 subjects: 55 patients after surgical treatment of acetabular fracture - the study population (mean age 43.6 ± 14.8 years) and 55 healthy subjects - the clinical control group (mean age 43.8 ± 14.9 years).

To ensure reliability of results, controls were individually matched to appropriate study population patients, in terms age, sex, body height and mass.

The study was conducted in Public Hospital and the protocol was approved by the Commission of Ethics (SKE 01-21/2014).

Investigators measured static balance in double leg stance (eyes open/eyes closed) for 30s on CQStab2P, a double module stabilometric platform.

The pain component of the Harris Hip score and the quality of fracture reduction (according to Matta's criteria) in digitized anteroposterior and two oblique view radiographs were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate in the study,
* full legal age,
* surgically treated hip acetabular fracture,
* time after the surgery between 3 and 84 months,
* full cognitive abilities, -full medical documentation, - the ability to fully load the operated limb (doctor's consent).

Exclusion Criteria:

* craniocerebral injuries,
* visual system disorders,
* neurological disorders,
* ear and sinuses infections,
* spinal pain
* injuries to the lower extremities,
* chronic illnesses (cancer, Parkinson's disease, epilepsy, diabetes, neuro-muscular disorders, uncontrolled coronary heart disease),
* taking psychoactive substances,
* lower limb thrombosis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population involved 55 patients after surgical treatment of hip acetabular fracture.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Static balance assessment with eyes open and closed | 2014-2017
  Static balance parameters were analysed.

SECONDARY OUTCOMES:
Harris hip score | 2014-2017
  Investigators determined patients' functional state on the basis of Harris Hip Score (HPP). This is an orthopedic tool which assesses functional state of patients after hip interventions. Harris hip score showed high validity and reliability. The tool assesses the following aspects: pain in the operated limb, hip movement range (registered with hand held goniometer), gait (limp, the distance a patient is able to walk, using mobility aids), other activities (walking the stairs, putting on shoes, and sitting, using public transport). Patients scored points for each analyzed element. The maximum number of points was 100. The score reflected the level of patient's functional state (a greater number of points meant that the patient had better ability). Then, we compared the results to the norms.
Merle d'aubigné score | 2014-2017
  disability score
Body mass index | 2014-2017
  Body weight and height will be collected

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aprato A, Joeris A, Tosto F, Kalampoki V, Stucchi A, Masse A. Direct and indirect costs of surgically treated pelvic fractures. Arch Orthop Trauma Surg. 2016 Mar;136(3):325-30. doi: 10.1007/s00402-015-2373-9. Epub 2015 Dec 11. PMID 26660303
- [Background] Arokoski JP, Leinonen V, Arokoski MH, Aalto H, Valtonen H. Postural control in male patients with hip osteoarthritis. Gait Posture. 2006 Jan;23(1):45-50. doi: 10.1016/j.gaitpost.2004.11.017. Epub 2005 Jan 18. PMID 16311194
- [Background] Bhat NA, Kangoo KA, Wani IH, Wali GR, Muzaffar N, Dar RA. Operative management of displaced acetabular fractures: an institutional experience with a midterm follow-up. Ortop Traumatol Rehabil. 2014 May-Jun;16(3):245-52. doi: 10.5604/15093492.1112281. PMID 25058100
- [Background] Baschera D, Rad H, Collopy D, Zellweger R. Incidence and clinical relevance of heterotopic ossification after internal fixation of acetabular fractures: retrospective cohort and case control study. J Orthop Surg Res. 2015 May 9;10:60. doi: 10.1186/s13018-015-0202-z. PMID 25956896
- [Background] Edgren J, Salpakoski A, Rantanen T, Heinonen A, Kallinen M, von Bonsdorff MB, Portegijs E, Sihvonen S, Sipila S. Balance confidence and functional balance are associated with physical disability after hip fracture. Gait Posture. 2013 Feb;37(2):201-5. doi: 10.1016/j.gaitpost.2012.07.001. Epub 2012 Aug 9. PMID 22884315
- [Derived] Dadura E, Truszczynska-Baszak A, Szydlowski D. Radiological and Functional Assessment of Treatment Outcomes in Patients after Open Reduction with Internal Fixation (ORIF) of Acetabular Fractures. Int J Environ Res Public Health. 2022 Jan 24;19(3):1277. doi: 10.3390/ijerph19031277. PMID 35162298